CLINICAL TRIAL: NCT04428008
Title: A Pilot Trial of Thymalfasin (Ta1) to Prevent COVID-19 Infection in Renal Dialysis Patients
Brief Title: Thymosin Alpha 1 to Prevent COVID-19 Infection in Renal Dialysis Patients
Acronym: Ta1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: William B. Ershler, MD (Other)
Collaborators: Davita Clinical Research (Industry); Ahmed Awad, MD (Unknown)
Responsible Party: Sponsor-Investigator, William B. Ershler, MD, Hematology Consultant (Private), Ershler, William B., MD
Organization: Ershler, William B., MD (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACW-1221958-1
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: COVID-19
Keywords: COVID-19; Thymalfasin; Thymosin alpha 1; ZADAXIN; Hemodialysis
MeSH Terms: conditions — COVID-19 | interventions — Thymalfasin; Trace amine-associated receptor 1

STUDY DESIGN:
Intervention Model Description: Subjects will be centrally randomized to receive either study treatment drug (Ta1) or no Ta1. Randomization will be stratified by site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active arm (Experimental): 1.6 mg thymalfasin in 1 mL subcutaneous injection twice weekly after dialysis for 8 weeks
  Interventions: Drug: Thymalfasin
- Control arm (No Intervention): Standard care

INTERVENTIONS:
Drug: Thymalfasin — Synthetic 28 amino acid peptide
  Other Names: Thymosin alpha 1; Ta1; ZADAXIN
  Arms: Active arm

SUMMARY:
Thymalfasin (thymosin alpha 1 or Ta1), the active pharmaceutical ingredient in ZADAXIN® injection, is a 28-amino acid synthetic peptide, identical to natural Ta1 produced by the thymus gland. Ta1 is a biological response modifier which activates various cells of the immune system, and is therefore expected to have clinical benefits in disorders where immune responses are impaired or ineffective, including acute and chronic viral and bacterial infections, cancers, and vaccine non-responsiveness. Patients with end-stage renal disease (ESRD) on hemodialysis, in addition to their intrinsic kidney disease and frequent burden of comorbidities, also have increased risk of exposure to communicable diseases as they are treated several times each week at hemodialysis centers with several other patients and clinic staff in attendance. The majority of patients are over 60 years of age and many are receiving immunosuppressive medications. Accordingly, ESRD patients are particularly susceptible to COVID-19 infection. Ta1 has been shown to be safely administered to hemodialysis patients. It is our hypothesis that a course of Ta1 administered to individuals with ESRD will reduce the rate and severity of infection with COVID-19.

DETAILED DESCRIPTION:
Patients with end-stage renal disease (ESRD) on hemodialysis, in addition to their intrinsic kidney disease and frequent burden of comorbidities, also have increased risk of exposure to communicable diseases as they are treated several times each week at hemodialysis centers with several other patients and clinic staff in attendance. The majority of patients are over 60 years of age and many are receiving immunosuppressive medications. Accordingly, ESRD patients are particularly susceptible to COVID-19 infection.

Thymalfasin (thymosin alpha 1, Ta1) is a naturally occurring peptide that has been evaluated for its immunomodulatory activities and related therapeutic potential in several conditions and diseases, including infectious disease and cancer. ZADAXIN, a synthetic form of Ta1, been has been used clinically in pilot studies for treatment of severe acute respiratory syndrome (SARS) and other lung infections including acute respiratory distress syndrome (ARDS) and chronic obstructive pulmonary disorder (COPD), as well as infections after bone marrow transplant]. Larger clinical trials have shown significant efficacy for treatment of severe sepsis and hepatitis B, along with certain cancers such as melanoma, hepatocellular, and lung cancer. Ta1 has also demonstrated improvement in response to vaccines in the elderly and in patients immunocompromised by renal disease. The beneficial clinical effects of Ta1 result from activation of toll-like receptor (TLR) 9 in dendritic and other immune system cells, resulting in augmentation of T helper (Th1) function, natural killer (NK) cell activity, and increased antibody responses to T-cell dependent antigens. Importantly, Ta1 also leads to an increase in IL-10 producing regulatory T cells, which create feedback inhibition of cytokine production, hence dampening immune response and preventing a pro-inflammatory cytokine storm.

It is our hypothesis that a course of Ta1 administered to individuals at high risk for COVID-19 infection (hemodialysis patients) will reduce the rate of COVID-19 infection and severity of infection with COVID-19, compared to untreated individuals in the same hemodialysis units with comparable risk. The study will also evaluate the need for hospitalization in those patients who do not become infected with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Signed informed consent
* End-stage renal disease (ESRD) who receive hemodialysis 2 or more times each week and are expected to continue on dialysis indefinitely.

Exclusion Criteria:

* Patients on short-term hemodialysis, such as those with transient renal dysfunction associated with acute illness who are projected to have return in renal function
* Patients for whom renal transplantation is anticipated within the next six months
* Patients with an anticipated survival of less than 3 months
* Patients with symptoms that might be attributable to COVID-19 infection
* Patients who test positive for SARS-CoV2
* Patients with active infectious disease requiring antibiotics
* Patients with hospitalization within the previous 3 months for acute myocardial infarction or congestive heart failure
* Patients with advanced malignancy receiving cytotoxic chemotherapy
* Patients with a Karnofsky Performance Scale score of less than 60
* Patients with prior history of solid organ (kidney, liver, heart, lung, pancreas) or bone marrow transplant
* Patients with active autoimmune disease on immunosuppressive medication
* Patients receiving Plaquenil
* Participation in an investigational drug or device trial in previous 30 days
* History of allergy or intolerance to Ta1
* Any other medical or psychiatric condition that, in the opinion of the Investigator, would compromise patient safety or interfere with the objectives of the protocol or completion of the protocol treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Reduction in documented infection with COVID-19 Reduction in infection with COVID-19 | 6 months
  Number of subjects who become infected with COVID-19 over the course of the study

SECONDARY OUTCOMES:
Need for hospitalization | 6 months
  Number of subjects who become hospitalized
Hospital length of stay | 6 months
  If subject becomes hospitalized, what length of time does the subject remain hospitalized
Need for ICU admission | 6 months
  Number of subjects who are entered into the ICU
ICU length of stay | 6 months
  If subject is entered into the ICU, what length of time does the subject remain in the ICU
Need for mechanical ventilation | 6 months
  Number of subjects who require mechanical ventilation
Duration of mechanical ventilation | 6 months
  If mechanical ventilation is required, what length of time the ventilation is required
Recovery time from COVID-19 | 6 months
  If subject becomes infected with COVID-19, how long does the subject require to recover from the infection
Change in any existing comorbidities or occurrence of newly diagnosed disease | 6 months
  Evaluation of whether any comorbidities are changed over the course of treatment (eg., worsening of congestive heart failure)
Incidence of non-COVID-19 infections | 6 months
  Determination of whether there are more or fewer infections other than COVID-19 (other respiratory, urinary tract, cellulitis, etc.)
Change in lymphocyte subsets (CD4, CD8) | 6 months
  Evaluation of the levels of CD4 and CD8 subjects
Mortality | 6 months
  Number of subjects who die during the course of the study
Treatment-emergent adverse events | 6 months
  Number of subjects with mild, moderate, or severe adverse events based on perceived clinical significance of the event
Treatment-emergent changes in vital signs | 6 months
  Number of subjects with mild, moderate, or severe changes to vital signs based on perceived clinical significance of the event
Treatment-emergent laboratory parameters | 6 months
  Number of subjects with mild, moderate, or severe laboratory findings based on perceived clinical significance of the event

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Consultants, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No